CLINICAL TRIAL: NCT03405831
Title: The Effect of Ivabradine Treatment on Exercise Capacity in Patients With Cardiac Allograft Vasculopathy After Heart Transplantation
Brief Title: Effect of Ivabradine on Exercise Capacity After Heart Transplantation
Acronym: VANISH-CAV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Finn Gustafsson (Other)
Collaborators: Danish Heart Foundation (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, MD, PhD, DMSci; Professor of Cardiology; Team Leader Advanced Heart Failure, Transplantation and Mechanical Circulatory Support; Department of Cardiology; The Heart Center; Copenhagen University Hospital; Rigshospitalet, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-HJE-LN-01
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Allograft Vasculopathy; Transplanted Heart Complication
Keywords: Heart transplantation; Exercise capacity; Heart rate; Cardiac allograft vasculopathy
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: This is a prospective single-center, double-blinded, placebo controlled, randomized study in long-term heart transplant recipients.
  Patients who meet the eligibility criteria will be randomized 1:1 at inclusion for one of two treatment groups: (i) treatment with ivabradine 5 mg bid or (ii) treatment with placebo bid for a period of 12 weeks. 35 participants will be enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine (Active Comparator): Study participants in this arm will receive ivabradin 5 mg bid for a period of 12 weeks.
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator): Study participants in this arm will receive placebo bid for a period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Ivabradine, oral tablets, 5 mg, coated in gelatine capsules to ensure blinding, 1 capsule twice a day, for a period of 12 weeks
  Other Names: Procoralan
  Arms: Ivabradine
Drug: Placebo — Placebo, gelatine capsules to ensure blinding, 1 capsule twice daily, for a period of 12 weeks
  Arms: Placebo

SUMMARY:
This study evaluates whether treatment with ivabradine compared to placebo can improve exercise capacity in long-term heart transplant recipients with cardiac allograft vasculopathy and elevated heart rate at rest.

Patients will receive treatment with either ivabradin or placebo for a period of 12 weeks.

DETAILED DESCRIPTION:
Elevated resting heart rate (HR) is a normal finding after successful heart transplantation (HTx) due to parasympathetic denervation at the operation.

Elevated resting HR is generally acknowledged as a negative predictor of outcome in heart disease. The impact in heart transplant recipients is not fully understood, however, it has been associated with increased risk of developing cardiac allograft vasculopathy (CAV) or death.

Cardiac allograft vasculopathy is a diffuse vascular disease affecting the entire coronary tree. It is the leading cause of death in patients more than 5 years after HTx and it is well known that patients with CAV have markedly reduced exercise capacity.

The association between elevated HR and CAV raises the question whether an intervention to specifically lower HR could improve symptoms and prognosis in heart transplant recipients with CAV and elevated resting HR.

Small studies have shown that HR reduction using the If channel blocker ivabradine after HTx is safe. However, none of these studies were randomized or blinded, and as such proof of any efficacy (beyond HR reduction) after HTx is non-existing. Clearly, there is a need to determine if such treatment could improve exercise capacity, graft function and prognosis after HTx.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 1 year post heart transplantation
* CAV verified by coronary angiography or intravascular ultrasound
* Resting HR > 80 bpm
* Age > 18 years
* Signed informed consent

Women, who have not yet entered menopause (defined as no menstrual bleeding in the last 12 months), will be required to provide a negative urine human chorionic gonadotropin (hCG) before entering the study and must use a safe birth control method in the total study period.

Exclusion Criteria:

* Rejection (>H1R) < 3 months
* Severe renal failure (estimated glomerular filtration rate (GFR) < 30 mL/min/1.73 m2)
* Inability or contraindication to perform a VO2 max test
* Presence of any condition that might per se influence exercise performance
* Known contraindication for treatment with ivabradine
* Hypersensitivity to the active substance or to any of the excipients of either study drug

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
ΔVO2max | The VO2max is assessed at baseline and 12 weeks follow-up.
  The change in VO2max (ΔVO2max) (mL/kg/min) from baseline to 12 weeks follow-up. The peak oxygen uptake (VO2max) reflects the maximal ability of a person to take in, transport and use oxygen, and it defines the functional aerobic capacity. It is used to provide an overall assessment of exercise capacity.

SECONDARY OUTCOMES:
ΔHRrest | 12 weeks
  Change in resting HR (beats/min) from baseline to 12 weeks follow-up
ΔHRreserve | 12 weeks
  Change in HR reserve (beats/min) from baseline to 12 weeks follow-up
ΔLVmass | 12 weeks
  Change in left ventricular (LV) mass (g) evaluated by cardiac MRI from baseline to 12 weeks follow-up
ΔLVEF | 12 weeks
  Change in left ventricular ejection fraction (LVEF) (%) evaluated by cardiac MRI from baseline to 12 weeks follow-up
Δmitral deceleration time | 12 weeks
  Change in mitral decelaration time (ms) evaluated by echocardiography from baseline to 12 weeks follow-up
ΔE/é | 12 weeks
  Change in E/é evaluated by echocardiography from baseline to 12 weeks follow-up
ΔE/A ratio | 12 weeks
  Change in E/A ratio evaluated by echocardiography from baseline to 12 weeks follow-up
Δisovolumetric relaxation time | 12 weeks
  Change in isovolumetric relaxation time (ms) evaluated by echocardiography from baseline to 12 weeks follow-up
Δtransmitral flow rate | 12 weeks
  Change in transmitral flow rate (volume/min) evaluated by cardiac MRI from baseline to 12 weeks follow-up
Δpulmonary venous flow | 12 weeks
  Change in pulmonary venous flow (volume/min) evaluated by cardiac MRI from baseline to 12 weeks follow-up
ΔLVEDV | 12 weeks
  Change in LVEDV (left ventricular end diastolic volume) (ml) evaluated by cardiac MRI from baseline to 12 weeks follow-up
ΔLVESV | 12 weeks
  Change in LVESV (left ventricular end systolic volume) (ml) evaluated by cardiac MRI from baseline to 12 weeks follow-up
ΔLV peak filling rate | 12 weeks
  Change in left ventricular (LV) peak filling rate (volume/min) evaluated by cardiac MRI from baseline to 12 weeks follow-up
Δtime to peak filling | 12 weeks
  Change in time to peak filling (sec) evaluated by cardiac MRI from baseline to 12 weeks follow-up
ΔQOL KCCQ | 12 weeks
  Change in QOL score evaluated by Kansas City Cardiomyopathy Questionnaire from baseline to 12 weeks follow-up
ΔQOL EQ-5D-5L | 12 weeks
  Change in QOL score evaluated by EQ-5D-5L questionnaire from baseline to 12 weeks follow-up

OTHER OUTCOMES:
Coronary vessel characterization | Substudy objective is only evaluated at baseline
  Substudy objective: To characterize coronary vessels in CAV using new imaging modalities and relating them to functional parameters of cardiac function. Modalities performed at baseline: Intravascular ultrasound (IVUS)/Near-infrared spectroscopy (NIRS), optical coherence tomography (OCT), 82-Rubudium positron emission tomography (PET) scan

CONTACTS AND LOCATIONS:
Overall Officials: Lærke Nelson, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiology, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No